CLINICAL TRIAL: NCT03171701
Title: Role of Color Doppler Ultrasonography in Prediction of Arteriovenous Fistula Maturation and Its Complications in Hemodialysis Patients
Brief Title: Color Doppler Ultrasonography in Prediction of Arteriovenous Fistula Maturation in Hemodialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, HFoad, Hadil Mohamed, Assiut University
Other Study IDs: arteriovenous fistula
Record Dates: First submitted 2017-05-29; First posted 2017-05-31 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Arteriovenous Fistula
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- maturation of arteriovenous fistula

SUMMARY:
The transplant is the definitive treatment of renal insufficiency, in our days. While waiting for it, the arteriovenous fistula surgery is standard procedure.

DETAILED DESCRIPTION:
Ultrasound is the main method of diagnostic imaging, because of its low cost, noninvasive without ionizing radiation associated or iodized contrast.

Vascular procedures and their complications represent a major cause of morbidity hospitalization and cost for patients in hemodialysis .

Many fistulas do not mature appropriately for being used in dialysis. So,The early recognition through the ultrasound examination of problems in the arteriovenous fistula maturation or possible complications that may compromise their viability, offers the opportunity of correction or appropriate treatment .

Criteria for maturation after arteriovenous fistula creation:

* Vein diameter larger than 4 mm remote from the site of fistula.
* Vein located at a depth of <5 mm from skin surface.

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients Of Chronic Renal Failure With Newly Placed AVF. 2)Clinically Stable Patients For Assessment Of Maturation Of AVF. 3) Complaints Of Hand Pain Or Numbness Following Creation Of The Access.

Exclusion Criteria:

* 1)Previously Failed AV Fistulas. 2)Deformed Or Scarred Upper Limb.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will be performed at Radiodiagnostic department, Assiut Police Hospital and assiut university hospital on all newly placed arteriovenous fistula for hemodialysis.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2018-07-01 (Estimated); Study Completion 2018-10-01 (Estimated)

PRIMARY OUTCOMES:
Role of color Doppler ultrasonography in prediction of arteriovenous fistula maturation and its complications in hemodialysis patients | one month
  Assess and monitor the maturation of the newly placed Arteriovenous fistulas, and to provide timely interventions for AV fistulas which are failing to mature

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malovrh M. Postoperative assessment of vascular access. J Vasc Access. 2014;15 Suppl 7:S10-4. doi: 10.5301/jva.5000243. Epub 2014 Apr 17. PMID 24817448